CLINICAL TRIAL: NCT04867564
Title: Radiation-induced Cardiac Toxicity After Non-small Cell Lung Cancer Radiotherapy Detected by Speckle-tracking Echocardiography
Brief Title: Radiation-induced Cardiac Toxicity After Non-small Cell Lung Cancer Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Joanna Socha, Principal Investigator, Military Institute od Medicine National Research Institute
Other Study IDs: 20/WIM/2021
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Non-small Cell Lung Cancer; Radiation Toxicity; Cardiac Toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Injuries; Cardiotoxicity | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients treated with curative radiotherapy: Consecutive NSCLC patients treated with standard RT with curative intent with or without platinum-based CHT
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Traditional echocardiography and speckle tracking echocardiography (STE) before and 1, 6, and 12 months after RT

SUMMARY:
Despite the growing interest in investigating how the radiotherapy (RT) dose to anatomical substructures of the heart links to survival, the heart substructures at risk remain poorly defined. They are not delineated routinely as part of the RT planning process and there is no consensus on their dose constrains. With improving prognosis for non-small cell lung cancer (NSCLC) patients, the evidence relating irradiation of the heart to excess mortality has begun to accumulate.

The study aims to evaluate subclinical cardiac dysfunction in consecutive NSCLC patients treated with definitive RT and to investigate the predictive value of the heart substructures dosimetric parameters for subclinical and overt cardiac toxicity as assessed using traditional and speckle tracking echocardiography (STE). The study will also investigate whether subclinical alterations detected by echocardiography with strain imaging may serve as a marker for future clinical dysfunctions.

DETAILED DESCRIPTION:
BACKGROUND Radiation-induced cardiac toxicity after RT for breast cancer or haematological malignancies is well described, with various studies linking post-RT cardiac morbidity and mortality with radiation dose. In patients treated with RT for NSCLC the associated heart exposure is higher than in breast cancer patients, and may lead to side effects possibly reducing survival. With improving prognosis for these patients after RT, the evidence began to accumulate that overall survival (OS) after RT for NSCLC is related to the heart dose. A landmark randomized trial Radiation Therapy Oncology Group (RTOG) 0617 failed to show any OS benefit with higher RT dose, and a post-hoc analysis revealed that the heart dose was a strong predictor of inferior OS. However, heart doses are higher with lower lobe tumors irradiation where irradiated volumes are larger due to respiratory tumor motion, and better blood supply of these parts of the lungs makes the lung toxicity worse, which also affects survival. Moreover, higher heart doses result from larger target volumes, which are themselves associated with worse OS. Therefore, a prospective evaluation of the cardiac toxicity after RT for NSCLC is needed to determine whether there is a correlation between the RT dose and specific types of cardiotoxicities.

Cardiac toxicity may manifest as any of a broad spectrum of diseases: as congestive heart failure, coronary ischemia, arrythmias or conduction abnormalities, and valvular and pericardial disease, therefore it is important to evaluate dosimetric parameters of the cardiac substructures, and to correlate them with potential adverse effects. Retrospective data suggests that the predictive value for cardiac events of the doses for the corresponding heart substructures outperforms the whole heart doses. STE is a valuable tool for a quantitative analysis of the changes to the cardiac substructures. Global longitudinal strain (GLS) has been regarded as a more accurate and sensitive parameter than left ventricle ejection fraction in assessing cardiac dysfunction, and its utility in the identification of subclinical myocardial changes has been demonstrated in a variety of conditions, including hypertension, diabetes mellitus, Cushing's disease, and chemotherapy- and RT-related cardiotoxicity. Recently, GLS has also been proved useful in the evaluation of the function of both atria and a right ventricle. Thus, STE is a non-invasive method allowing not only for the identification but also for the quantitative evaluation of subclinical systolic dysfunction of all the heart chambers.

In the present study, subclinical myocardial dysfunction will be evaluated using STE before and 1, 6, and 12 months after RT in consecutive NSCLC patients treated with definitive RT with or without chemotherapy (CHT) and the association between early cardiac effects and RT dose distribution in the corresponding heart substructures will be explored. Moreover, the study will show whether subclinical alterations detected by strain imaging precede the occurrence of clinical dysfunctions, possibly allowing for earlier treatment or closer monitoring of such patients.

OBJECTIVES OF THE STUDY The aim of this prospective study is to evaluate subclinical cardiac dysfunction in consecutive NSCLC patients treated with definitive RT and to investigate the predictive value of the cardiac substructures dosimetric parameters for cardiac toxicity as evaluated using STE and traditional echocardiographic parameters. The study will also investigate whether subclinical alterations detected by echocardiography with strain imaging may serve as a marker for future clinical dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to provide informed consent
* Histologically confirmed non-small cell carcinoma of the lung
* Patient to receive standard RT with curative intent with or without concurrent or sequential CHT according to the institutional protocol
* ECOG performance status 0-1 within one month of accrual
* Negative pregnancy test within one month of accrual if woman is premenopausal
* Patient presented at multidisciplinary tumor board or quality-assurance rounds
* Satisfactory pulmonary function tests, i.e., forced expiratory volume during the first second (FEV1) ≥ 1.0 l (≥40%)

Exclusion Criteria:

* Noncompliance with any of the inclusion criteria
* Pregnancy
* Prior RT to the thorax
* Patient to receive stereotactic body radiation therapy (SBRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in one institution (Military Institute of Medicine, Warsaw, Poland). Accrual of 50 patients a year is anticipated, the planned accrual period is two years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
RT-induced systolic and diastolic function alterations | 1 year
  Systolic and diastolic function alterations assessed using traditional echocardiographic parameters as well as speckle tracking echocardiography analysis at 1, 6, and 12 months after RT compared to baseline.

SECONDARY OUTCOMES:
The predictive value of cardiac substructures dosimetric parameters for cardiac toxicity as evaluated using STE and traditional echocardiographic parameters | 1 year
  Apart from the whole heart, which is routinely contoured, the following substructures will be also contoured on the computed tomography planning CT scans: left ventricle (LV), left ventricle anterior segment (LVant), left ventricle inferior segment (LVinf), left ventricle lateral segment (LVlat), left ventricle septal segment (LVsept), left atrium (LA), right ventricle (RV), right atrium (RA), aortic valve (AV), pulmonic valve (PV), tricuspid valve (TV), mitral valve (MV), left main coronary artery (LMCA), left anterior descending coronary artery (LAD), left circumflex coronary artery (LCxCA), and right coronary artery (RCA). No prespecified dose constrains will be applied for these substructures. RT treatment plan will be prepared using routine whole heart dose constrains according to the institutional protocol, and the pre-specified dose-volume histogram parameters will be extracted for analysis.
The predictive value of subclinical alterations detected by echocardiography for future clinical dysfunctions | 1 year
  Occurence of the symptomatic cardiac disorders, as classified by Common Terminology Criteria for Adverse Events (CTCAE) v.4.0, in patients with vs. without subclinical alterations detected by echocardiography
Cumulative incidence of cardiac disorders, as classified by CTCAE4.0 | 1 year
  Cumulative incidence of cardiac disorders, as classified by CTCAE4.0

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Socha, MD, PhD, Principal Investigator — Military Institute od Medicine National Research Institute
Locations (1):
- Department of Radiotherapy, Military Institute of Medicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The study data will be available following publication on request. Requests to: jsocha@wim.mil.pl